CLINICAL TRIAL: NCT01867866
Title: A Phase 1, Open-Label, Randomized, Parallel Group Study Evaluating the Pharmacokinetics of FTD as a Component of TAS-102 Compared With FTD Alone
Brief Title: Study Comparing the Pharmacokinetics of FTD as a Component of TAS-102 With FTD Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPU-TAS-102-102
Record Dates: First submitted 2013-05-24; First posted 2013-06-04 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors (excluding breast cancer) for which no standard therapy exists
MeSH Terms: interventions — trifluridine tipiracil drug combination; Trifluridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAS-102 (Experimental)
  Interventions: Drug: TAS-102
- FTD (Trifluridine) (Experimental)
  Interventions: Drug: Trifluridine

INTERVENTIONS:
Drug: TAS-102 — 35 mg/m2/dose, orally, twice daily on days 1-5 and 8-12 of each 28-day cycle. Number of cycles: until at least one of the discontinuation criteria is met.
  Arms: TAS-102
Drug: Trifluridine — 35 mg/m2, orally, single dose
  Arms: FTD (Trifluridine)

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of trifluorothymidine (FTD) as a component of TAS-102 with FTD alone.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, randomized, parallel, 2-group study evaluating the PK of FTD as a TAS-102 component compared with FTD alone in patients with advanced solid tumors (excluding breast cancer). Patients will be randomized to receive a single dose of TAS-102 or FTD during the PK contribution phase and will receive continuing cycles of TAS-102 during the extension phase.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Has advanced solid tumors (excluding breast cancer) for which no standard therapy exists
3. ECOG performance status of 0 or 1
4. Is able to take medications orally
5. Has adequate organ function (bone marrow, kidney and liver)
6. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion Criteria:

1. Has had certain other recent treatment e.g. anticancer therapy, received investigational agent, within the specified time frames prior to study drug administration
2. Certain serious illnesses or medical condition(s)
3. Has had either partial or total gastrectomy
4. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies
5. Known sensitivity to TAS-102 or its components
6. Is a pregnant or lactating female
7. Refuses to use an adequate means of contraception (including male patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
FTD pharmacokinetic parameters AUC0-last and Cmax | Day 1 of Cycle 1

SECONDARY OUTCOMES:
FTD pharmacokinetic parameters AUC0-inf, Tmax, T1/2, CL/F, and Vd/F | Day 1 of Cycle 1
FTY and TPI pharmacokinetic parameters AUC0-last, Cmax, AUC0-inf, Tmax, T1/2, CL/F, and Vd/F | Day 1 of Cycle 1
Multiple-dose FTD, FTY, and TPI pharmacokinetic parameters AUC0-last, Cmax, Tmax, T1/2 | Day 12 of Cycles 1, 2, and 3
Tumor assessments using Response Evaluation Criteria in Solid Tumors (RECIST) | Every 8 weeks through Cycle 6 (ie, through 24 weeks). Thereafter, assessments will be performed at least every 12 weeks according to site standard of care, until at least one of the treatment discontinuation criteria is met.
Safety monitoring including adverse events, vital signs, and laboratory assessments | Through 30 days following last administration of study medication or until initiation of new anticancer treatment
  Standard safety monitoring and grading using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Drew Rasco, MD, Principal Investigator — South Texas Accelerated Research Therapeutics, LLC
Locations (1):
- South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas, United States